CLINICAL TRIAL: NCT00003150
Title: Phase III Trial of CHOP Versus CHOP and Chimeric Anti-CD20 Monoclonal Antibody (IDEC-C2B8) in Older Patients With Diffuse Mixed, Diffuse Large Cell and Immunoblastic Large Cell Histology Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy With or Without Monoclonal Antibody Therapy in Treating Older Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); SWOG Cancer Research Network (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065935; ECOG-E4494; CLB-9793; SWOG-E4494
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2010-08

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — Rituximab; VAP-cyclo protocol; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

INTERVENTIONS:
Biological: rituximab
Drug: CHOP regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known if combination chemotherapy is more effective with or without rituximab for non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without rituximab in treating older patients who have non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of CHOP (cyclophosphamide, doxorubicin, vincristine, and prednisone) with or without rituximab in older patients with diffuse mixed, diffuse large, or immunoblastic large cell non-Hodgkin's lymphoma of B-cell lineage with respect to the response rate, time to treatment failure, toxicity, and survival. II. Compare the efficacy of maintenance therapy consisting of rituximab vs observation alone after initial therapy with respect to the time to treatment failure, duration of response, toxicity, and survival of this patient population. III. Determine if maintenance therapy with rituximab results in the conversion of any partial response to complete response.

OUTLINE: This is a randomized study. For the first randomization, patients are stratified according to the number of risk factors (0-1 vs 2-4). For the second randomization, in addition to the number of risk factors, patients are stratified according to objective response to initial induction therapy (partial response vs complete response) and induction therapy (CHOP vs CHOP and rituximab). Patients are randomized to one of two treatment arms. Arm I: Patients receive CHOP chemotherapy comprising cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Treatment repeats every 21 days in the absence of unacceptable toxicity. Arm II: Patients receive treatment as in arm I. Patients also receive rituximab IV on days -7,-3, 41, and 83. Patients who achieve complete response (CR) after 4 courses of CHOP and remain in CR after 6 courses of CHOP are further randomized to one of two arms. Arm I (Maintenance therapy): Patients receive rituximab IV weekly for 4 weeks. Courses repeat every 6 months for 2 years in the absence of unacceptable toxicity. Arm II: Patients are observed. Patients who achieve partial response (PR) after 6 courses OR PR after 4 courses and then CR after 6 courses receive 2 additional courses of CHOP therapy. Patients are then also randomized to receive either maintenance therapy or observation as above. Patients with stable disease or disease progression are removed from the study. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 630 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven intermediate or high grade B-cell non-Hodgkin's lymphoma (other than Burkitt's, non-Burkitt's, undifferentiated, or lymphoblastic lymphoma) B-cell non-Hodgkin's lymphoma positive for CD19 and/or CD20 by slide-based immunohistochemistry or flow cytometry No mantle cell or follicular lymphoma Measurable disease, defined by at least one of the following: Physical examination Radiographic findings of at least 2 dimensions Bidimensional measurable defect or mass measuring at least 2 cm in diameter on radionuclide or CT scan Enlarged spleen extending at least 2 cm below the costal margin provided that there is no other likely explanation besides lymphomatous involvement Enlarged liver extending at least 5 cm below the costal margin along with biopsy-proven lymphomatous hepatic involvement No history of transformed lymphoma No known posttransplantation lymphoproliferative disorder No CNS involvement CALGB patients 60-65 years of age must not be eligible for any other study of higher priority A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: See Disease Characteristics 60 and over Performance status: ECOG 0-3 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 (unless due to lymphoma) Platelet count greater than 100,000/mm3 (unless due to lymphoma) Hepatic: Bilirubin no greater than 3.0 mg/dL Renal: Creatinine less than 2.1 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No active heart disease including congestive heart failure, myocardial infarction within the past 3 months, or symptomatic ventricular arrhythmia LVEF at least 45% if prior history of heart disease exists Other: HIV negative No other malignancy within the past 5 years except squamous cell or basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No prior biologic response modifier therapy No prior immunotherapy No prior rituximab Chemotherapy: No prior cytotoxic chemotherapy No concurrent dexrazoxane Endocrine therapy: Prior corticosteroids allowed Radiotherapy: No prior radiotherapy No prior radioimmunotherapy Surgery: Not specified

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 1997-12; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. Habermann, MD, Study Chair — Mayo Clinic; Vicki A. Morrison, MD, Study Chair — Veterans Affairs Medical Center - Minneapolis; James K. Weick, MD, Study Chair — Hematology Oncology Associates of the Palm Beaches
Locations (91):
- United States (91):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Hematology Oncology Associates, Atlantis, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Advani RH, Chen H, Habermann TM, Morrison VA, Weller EA, Fisher RI, Peterson BA, Gascoyne RD, Horning SJ; Eastern Cooperative Oncology Group; Cancer and Leukemia Group B; Southwest Oncology Group. Comparison of conventional prognostic indices in patients older than 60 years with diffuse large B-cell lymphoma treated with R-CHOP in the US Intergroup Study (ECOG 4494, CALGB 9793): consideration of age greater than 70 years in an elderly prognostic index (E-IPI). Br J Haematol. 2010 Oct;151(2):143-51. doi: 10.1111/j.1365-2141.2010.08331.x. PMID 20735398
- [Result] Winter JN, Li S, Aurora V, Variakojis D, Nelson B, Krajewska M, Zhang L, Habermann TM, Fisher RI, Macon WR, Chhanabhai M, Felgar RE, Hsi ED, Medeiros LJ, Weick JK, Weller EA, Melnick A, Reed JC, Horning SJ, Gascoyne RD. Expression of p21 protein predicts clinical outcome in DLBCL patients older than 60 years treated with R-CHOP but not CHOP: a prospective ECOG and Southwest Oncology Group correlative study on E4494. Clin Cancer Res. 2010 Apr 15;16(8):2435-42. doi: 10.1158/1078-0432.CCR-09-1219. Epub 2010 Apr 6. PMID 20371683
- [Result] Aurora V, Li S, Horning SJ, et al.: Prognostic significance of p53/p21 expression in DLBCL treated with CHOP or R-CHOP: a correlative study of E4494. [Abstract] J Clin Oncol 25 (Suppl 18): A-8038, 450s, 2007.
- [Result] Morrison VA, Weller EA, Habermann TM, et al.: Maintenance rituximab (MR) compared to observation (OBS) after R-CHOP or CHOP in older patients (pts) with diffuse large B-cell lymphoma (DLBCL): an Intergroup E4494/C9793 update. [Abstract] J Clin Oncol 25 (Suppl 18): A-8011, 443s, 2007.
- [Result] Advani RH, Chen H, Habermann TM, et al.: Prognostic indices in older DLBCL patients receiving R-CHOP: an analysis of the U.S. Intergroup study (E4494, CALGB 9793). [Abstract] Blood 108 (11): A-813, 2006.
- [Result] Habermann TM, Weller EA, Morrison VA, Gascoyne RD, Cassileth PA, Cohn JB, Dakhil SR, Woda B, Fisher RI, Peterson BA, Horning SJ. Rituximab-CHOP versus CHOP alone or with maintenance rituximab in older patients with diffuse large B-cell lymphoma. J Clin Oncol. 2006 Jul 1;24(19):3121-7. doi: 10.1200/JCO.2005.05.1003. Epub 2006 Jun 5. PMID 16754935
- [Result] Winter JN, Weller EA, Horning SJ, Krajewska M, Variakojis D, Habermann TM, Fisher RI, Kurtin PJ, Macon WR, Chhanabhai M, Felgar RE, Hsi ED, Medeiros LJ, Weick JK, Reed JC, Gascoyne RD. Prognostic significance of Bcl-6 protein expression in DLBCL treated with CHOP or R-CHOP: a prospective correlative study. Blood. 2006 Jun 1;107(11):4207-13. doi: 10.1182/blood-2005-10-4222. Epub 2006 Jan 31. PMID 16449523
- [Result] Morrison V, Weller E, Habermann T, et al.: Dose intensity of CHOP alone or with rituximab in diffuse large B-cell lymphoma (DLBCL) in patients >60 years of age: an analysis of the intergroup trial ( CALGB 9793, ECOG-SWOG 4494). [Abstract] Ann Oncol 16 (Suppl 5): A-224, v102, 2005.
- [Result] Habermann TM, Weller E, Morrison VA, et al.: Rituximab-CHOP versus CHOP with or without maintenance rituximab in patients 60 years of age or older with diffuse large B-cell lymphoma (DLBCL): an update. [Abstract] Blood 104 (11): A-127, 2004.
- [Result] Morrison VA, Weller EA, Habermann TM, Li S, Fisher RI, Cheson BD, Peterson BA. Patterns of growth factor usage and febrile neutropenia among older patients with diffuse large B-cell non-Hodgkin lymphoma treated with CHOP or R-CHOP: the Intergroup experience (CALGB 9793; ECOG-SWOG 4494). Leuk Lymphoma. 2017 Aug;58(8):1814-1822. doi: 10.1080/10428194.2016.1265111. Epub 2016 Dec 14. PMID 27967294